CLINICAL TRIAL: NCT00728884
Title: Observational Study of Certain Prevail Implant System in Maxillary and Mandibular Regions
Brief Title: Study of Certain Prevail Implants Used to Treat All Types of Edentulism in the Maxilla and Mandible
Acronym: PrevailMulti
Status: Completed | Type: Observational
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 2406
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Partial Edentulism
Keywords: dental implants; Certain Prevail; multicenter; clinical study; partial edentulism; total edentulism; platform switching; single stage; early loading; crestal bone level; single tooth replacements; short or long fixed bridges; overdenture; fixed denture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This observational, prospective clinical study evaluates the performance of the Certain Prevail implant system to show potential crestal bone and soft tissue preservation following the crestal bone. It will also evaluate implant performance.

Study (null) hypothesis: The preservation of crestal bone for the Certain Prevail implants will be the same as that for standard non-platform switched implants from contemporaneous studies (historical controls).

DETAILED DESCRIPTION:
This is a prospective, observational study of patients with partial or complete edentulism treated with the Certain Prevail dental implants. Restorations will consist of single tooth replacements, short and long fixed bridges, and overdentures and full dentures. All implants are placed using a single stage approach and temporalization occurring after two months of healing (early loading). Each center will strive to enroll a total of 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and any race greater than 18 years of age
* patients for whom a decision has already been made to use dental implants for treating an existing dental condition specifically:

  1. dental implants restored as single tooth replacements, short and long fixed bridges, overdenture, or fixed full denture.
  2. a temporary healing abutment will be placed on implant during implant placement surgery (single stage procedure).
* patients must be physically able to tolerate conventional surgical and restorative procedures
* patients must agree to be evaluated for each study visit, especially the yearly follow-up visit

Exclusion Criteria:

* patients with active infection or severe inflammation in the areas intended for implant placement
* patients with a >10 cigarette per day smoking habit
* patients with uncontrolled diabetes mellitus
* patients with metabolic bone disease
* patients who have had treatment with therapeutic radiation to the head within the past 12 months
* patients in need of allogenic bone grafting at the site of the intended study implant for augmentation purposes. Grafting for treatment of dehiscence or fenestration must have occurred at least 8 weeks prior to implant placement surgery
* patients who are pregnant at the screening visit
* patients with evidence of severe para-functional habits such as bruxing or clenching
* patients with less than 6 weeks of healing time post tooth extraction at the intended treatment site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These will be patients who are otherwise seeking dental implant therapy and belong to the study centers' standard patient population.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lorenzoni, DMD, MD, PhD, Principal Investigator — MEDIZINISCHE UNIVERSITAT GRAZ
Locations (1):
- Medizinische Universitat Graz- Klinische Abteilung fur Zahnersatzkunde, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 200 patients will be enrolled across all participating centers, with enrollment efforts beginning in August 2005. Enrollment period remained until February 2007. Ten participating sites are private practices and two are Universities.
Pre-assignment Details: Pre-treatment included a screening visit (enroll those meeting all inclusion criteria),signing informed consent, and per-surgical data collection. Patients are then scheduled for implant placement surgery.
Groups:
- Certain Prevail Implants: Osseotite surfaced implants with internal connection
Period: Implant Placement Surgery
Arm/Group | Certain Prevail Implants
Started | 162
Completed | 162
Not Completed | 0
Period: Permanent Prosthesis Placement
Arm/Group | Certain Prevail Implants
Started | 162
Completed | 149
Not Completed | 13
Not completed — Lost to Follow-up | 13
Period: One Year Post Placement Follow-up
Arm/Group | Certain Prevail Implants
Started | 149
Completed | 145
Not Completed | 4
Not completed — Lost to Follow-up | 4
Period: Two Year Post Placement Follow-up
Arm/Group | Certain Prevail Implants
Started | 145
Completed | 145
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Certain Prevail Implants
Number analyzed (Participants) | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 63
Region of Enrollment [Number; unit: participants]
  Austria | 26
  Australia | 10
  Ireland | 14
  United States | 31
  Italy | 52
  France | 9
  Sweden | 20

OUTCOME MEASURES:

1. Primary Outcome: Osseous Integration
Time Frame: one year
Population: total number of patients enrolled in the study were analyzed at this time (patients with implants not showing mobility).Patients receiving study implant(s) will achieve integration success (implant show no signs of mobility) of the implant at the time of analysis.
Measure: Number; unit: participants
Arm/Group | Certain Prevail Implants
Number analyzed (Participants) | 162
participants | 145

2. Secondary Outcome: Crestal Bone Resorption
Description: Crestal bone level measures- changes from baseline to last study visit
Time Frame: four years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event reports are collected from day to present, 3 years study duration to date.
Description: Adverse event data is collected during each study event visit the patient is seen for.
Arm/Group | Certain Prevail Implants
Serious Adverse Events (participants affected / at risk) | 0/162
Other Adverse Events (participants affected / at risk) | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall furnish SPONSOR with a copy of any proposed publication thirty (30) days prior to submission for publication for review and comment. SPONSOR may request PI to delay publishing such proposed publication for a maximum of an additional sixty (60) days in order to protect the potential patentability of any invention described therein.